CLINICAL TRIAL: NCT01817881
Title: Investigation of the Accuracy in the Use of Temporal Artery Thermometers for Non-invasive Temperature Measurement
Brief Title: Investigation of the Accuracy of Temporal Artery Thermometers
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christian Maschmann, MD, MD, Bispebjerg Hospital
Other Study IDs: 2013-BBH-AKM/MMA-Exerg
Record Dates: First submitted 2013-03-18; First posted 2013-03-26 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether temporal artery thermometers are accurate tools in temperature measurements of patients presenting to the Emergency Department. The investigators´ hypothesis is that there is a difference of > 0,3 degrees centigrade (Bland-Altman) between the temperatures measured with the temporal artery thermometers used at the investigators´ hospital (Exergen TAT-5000) and those measured with rectal thermometers (OMRON MC-341-E), which is considered to be the gold standard in Denmark defined by the Danish Center for Clinical Guidelines. The investigators furthermore hypothesize that the difference between these measurements is greater if measured in a patient with hyperthermia (temperature > 37,9 degrees Centigrade).

DETAILED DESCRIPTION:
Accurate temperature measurement on patients presenting to the Emergency Department is of great importance since it has significant influence on the further treatment of the patient. At Bispebjerg Hospital temporal artery thermometers are being implemented as they provide a fast and comfortable temperature measurement compared to rectal thermometers, who are considered to be the gold standard, defined by the Danish Center for Clinical Guidelines. The scientific proof for their accuracy compared to rectal thermometers in adult patients is insufficient though. The purpose of this study is to determine the difference between temperatures measured by a temporal artery thermometer (Exergen TAT-5000) and a rectal thermometer (OMRON MC-341-E) in patients presenting to the Emergency Department at Copenhagen University Hospital: Bispebjerg. The investigators hypothesize that there will be an average difference of at least 0,3 degrees centigrade between those two types of measurements (Bland-Altman). Based on a significance of 5% and a power of 80% the number of patients was calculated to 385, including an estimated 10% dropout.

ELIGIBILITY:
Inclusion Criteria:

* given informed consent

Exclusion Criteria:

* constipation
* anal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Difference between temperatures measured by temporal artery thermometers and rectal thermometers | 6 months

SECONDARY OUTCOMES:
Reproducibility of temporal artery thermometers' measurements | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanne H Nygaard, RN, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Copenhagen University Hospital: Bispebjerg - AKM-MMA, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Nygaard H, Maschmann C, Ekmann A. Comparison between temporal and rectal temperature measurement. Dan Med J. 2020 Oct 20;67(11):A04200270. PMID 33215602